CLINICAL TRIAL: NCT05764590
Title: A Phase 2, Randomized, Open-Label, Active-Controlled, Multicenter Study to Evaluate the Safety and Serum Phosphorus Lowering Effect of AP-306 in Chronic Kidney Disease Patients Receiving Maintenance Hemodialysis With Hyperphosphatemia
Brief Title: A Study to Evaluate Safety and Efficacy of AP-306 in Hyperphosphatemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alebund Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP306-HP-01
Record Dates: First submitted 2023-02-17; First posted 2023-03-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Diseases; Hyperphosphatemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AP-306 (Experimental)
  Interventions: Drug: AP-306
- Sevelamer Carbonate (Active Comparator)
  Interventions: Drug: Sevelamer Carbonate

INTERVENTIONS:
Drug: AP-306 — A blood phosphorus lowering drug with a novel mechanism
  Arms: AP-306
Drug: Sevelamer Carbonate — A phosphate binder
  Arms: Sevelamer Carbonate

SUMMARY:
The goal of this clinical trial is to learn about the following questions in the patients receiving maintenance hemodialysis with elevated blood phosphorus:

* How much effect AP-306 has assessed by blood phosphorus lowering;
* How safe and tolerable AP-306 is.

Participants will receive either following treatments:

* AP-306, and
* Sevelamer carbonate.

ELIGIBILITY:
Important Inclusion Criteria:

1. On a stable hemodialysis regimen at a frequency of three times per week for at least 12 weeks prior to the screening visit
2. Dialysis sufficiency SpKt/V ≥ 1.2 at the screening visit or any documented result within 12 weeks prior to the screening visit
3. Serum phosphorus within the trial-required range

Important Exclusion Criteria:

1. Pregnant or breastfeeding
2. Any history of kidney transplant
3. Any history of a parathyroid intervention
4. Any clinically significant GI disorders within 4 weeks prior to the screening visit
5. Hospitalization for cardiac or cerebrovascular disease within 24 weeks prior to the screening visit
6. Hospitalization for cardiac or cerebrovascular disease within 24 weeks prior to the screening visit
7. Documented history of hypersensitivity or allergic reactions to any of the excipients used by AP-306, or history of hypersensitivity or allergic reactions or intolerant to sevelamer carbonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of AP-306 assessed by serum phosphorus lowering | 12 weeks
  The change in serum phosphorus level from the baseline to the end of treatment

OTHER OUTCOMES:
To evaluate the overall safety of AP-306 assessed by incidence of treatment-emergent adverse events | 15 weeks
  All adverse events occurred after the study treatment initiation will be collected and their nature, frequency, and severity will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Li Wang, MD, Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No